CLINICAL TRIAL: NCT03727828
Title: Diagnostic, Risk Stratification and Prognostic Value of Novel Biomarkers in Patients With Heart Failure: DRAGON-HF Study
Brief Title: Diagnostic, Risk Stratification and Prognostic Value of Novel Biomarkers in Patients With Heart Failure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Collaborators: Tongji Hospital (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Nanfang Hospital, Southern Medical University (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Chinese Academy of Medical Sciences, Fuwai Hospital (Other); Yangpu Hospital (Unknown); Shanghai Municipal Hospital of Traditional Chinese Medicine (Other); Huashan Hospital Baoshan Branch (Unknown); Shanghai Zhongye Hospital (Unknown); Shanghai BaoshanLuodianHospital (Unknown); Shanghai Shibei Hospital (Unknown); Nantong Sixth People's Hospital (Unknown)
Responsible Party: Principal Investigator, Ya-Wei Xu, Professor, Shanghai 10th People's Hospital
Other Study IDs: DRAGON-HF
Record Dates: First submitted 2018-10-21; First posted 2018-11-01 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood collected at various time points according to the study cohort.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with heart failure: Patients with heart failure (HF) who are followed in the hospital or clinic setting, with optimization of medical therapy and blood collection.
  Interventions: Diagnostic Test: Patients with heart failure
- healthy control

INTERVENTIONS:
Diagnostic Test: Patients with heart failure — Participants will have serial blood collection on medical therapy for heart failure
  Groups: Patients with heart failure

SUMMARY:
The objective of this work is to investigate and then to sequence new biomarkers in the blood of patients with heart failure, and study their diagnostic, risk stratification and prognostic value.

DETAILED DESCRIPTION:
Blood samples (plasma or serum) for heart failure patients presenting dyspnea or edema and with increased NT-proBNP. The objective of this work is to investigate and then to sequence new proteins or microRNAs in the blood of these patients for diagnostic, risk stratification and prognostic purpose.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years of age
2. Symptomatic (NYHA class II-IV) heart failure (as diagnosed by clinician, radiographic images, or abnormal natriuretic peptide level)
3. Hospital admission, Emergency Department visit, or outpatient diuretic escalation of therapy for destabilized HF at least once in the 6 months prior to enrollment

Exclusion Criteria:

1. Life expectancy <1 year due to causes other than HF such as advanced cancer
2. Cardiac transplantation or revascularization indicated or expected within 6 months
3. Severe obstructive or restrictive pulmonary disease, defined as a forced expiratory volume in 1 sec <1 L (when diagnosed as standard of care)
4. Subject unable or unwilling to provide written informed consent
5. Coronary revascularization (percutaneous coronary intervention or bypass surgery) within the previous 3 months
6. Progressive neurological disease
7. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with heart failure.Patients presenting with shortness of breathor edema and with increased NT-proBNP.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2018-11-15 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of participants with cardiaovascular death after 5-year follow up | 5 years
  The cardiovascular mortality after 5-year follow up will be assessed to detect prognostic values of circulating biomarkers
Time to decompensated heart failure (HF) requiring in-patient admission or ER visit or IV diuretic therapy in the outpatient realm | 5 years
  New onset of classic symptoms and signs of destabilized HF, including lower extremity edema, jugular venous distension, bibasilar crackles, orthopnea and paroxysmal nocturnal dyspnea.

SECONDARY OUTCOMES:
Comparison of new biomarker with NT-ProBNP on diagnostic value in patients with heart failure | 1 year
  Compare the sensitivity and specificity of new biomarker with NT-ProBNP to assess the accuracy of diagnostic value in discriminating heart failure from non-heart failure participants.
Change From Baseline in left ventricular ejection fraction | 5 years
  Assess the change in left ventricular ejection fraction at the end of 5-year follow up.
Change From Baseline in left ventricular end-systolic volume | 5 years
  Assess the change in left ventricular end-systolic volume at the end of 5-year follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Dachun Xu, Ph.D, Principal Investigator — Shanghai 10th People's Hospital
Locations (1):
- Shanghai Tenth People's Hospital, Tongji University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be available with reasonable request.

REFERENCES:
- [Derived] Wang Z, Zhu Z, Shen J, Zhang Y, Wang T, Xu Y, Jiang D, Liu W. Predictive value of remnant cholesterol for left ventricular hypertrophy and prognosis in hypertensive patients with heart failure: a prospective study. Lipids Health Dis. 2024 Sep 12;23(1):294. doi: 10.1186/s12944-024-02282-y. PMID 39267042
- [Derived] Ma T, Huang R, Xu Y, Lv Y, Liu Y, Pan X, Dong J, Gao D, Wang Z, Zhang F, Yan C, Ong SB, Su Y, Xu D. Plasma GAS6 predicts mortality risk in acute heart failure patients: insights from the DRAGON-HF trial. J Transl Med. 2023 Jan 12;21(1):21. doi: 10.1186/s12967-022-03859-w. PMID 36635690
- [Derived] Su Y, Sun Y, Tang Y, Li H, Wang X, Pan X, Liu W, Zhang X, Zhang F, Xu Y, Yan C, Ong SB, Xu D. Circulating miR-19b-3p as a Novel Prognostic Biomarker for Acute Heart Failure. J Am Heart Assoc. 2021 Oct 19;10(20):e022304. doi: 10.1161/JAHA.121.022304. Epub 2021 Oct 6. PMID 34612058